CLINICAL TRIAL: NCT04779073
Title: Evaluation of Physiotherapists' Knowledge Level of Cardiopulmonary Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rabia Tugba Kilic, assistant professor, Ankara Yildirim Beyazıt University
Other Study IDs: 2020-281
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: physiotherapist cardiopulmonary resuscitation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was planned to determine the physiotherapists' knowledge and qualifications of CPR, their beliefs about the use of CPR in an emergency, and their perception of CPR competence.

DETAILED DESCRIPTION:
Cardiopulmonary arrest is a sudden stop of breathing and circulation. Resuscitation is an effort to restore spontaneous heartbeat, respiration and brain functions .Although it is actually a standard algorithm, the approach to cardiopulmonary resuscitation can vary among practitioners.Resuscitation success; practitioner, the state of the arrested person,It depends on several factors such as the resources and equipment available.

The main issue in the success of the resuscitation; how quickly the scene can be reached and how effective CPR can be performed.Guidelines on CPR, including resuscitation information, are updated by the American Heart Association (AHA) and the European Resuscitation Council (ERC) in various time periods.Although there are some differences in resuscitation practices, the importance of early diagnosis and rapid intervention are emphasized in both guidelines. The shortest possible time for the patient to return to life after cardiac arrest Basic Life Support (TYD) and Advanced Life Support (ADS) should be initiated in the period.TYD is applied by non-professional but trained individuals without any material or medication. On the other hand, IDE is applied by a professional team of health professionals using the necessary materials and medicines. It is possible to encounter a cardiac arrest anywhere inside or outside the hospital.

The fact that healthcare workers have been trained on TYD and VBS is an important factor in increasing the chances of arrest cases to come back to life.

Only two published studies on the attitudes of physiotherapists towards CPR have been identified in the literature. One of these was a study involving 140 hospital-based physiotherapists who investigated their knowledge, attitudes and practices in CPR in South-West Nigeria. The authors found that 64% of respondents had insufficient to average theoretical knowledge about CPR and only 45% of respondents held a positive attitude about the importance of CPR.

The second study was conducted with 2,614 healthcare professionals from two Swedish hospitals, where participants filled out a questionnaire about physical / mental discomfort and attitudes towards CPR before and after training. A total of 228 assistant health professionals were included in the sample, including physiotherapists, occupational therapists, psychologists, social workers, and biomedical analysts.

All healthcare professional groups relied more on CPR knowledge after training; however, one limitation of this is that they do not test pre- or post-practice CPR skills. Unfortunately, the applicability of the findings was limited, as the group of physiotherapists was an unidentified subset of 228 allied health professionals in the study.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists working in various institutions and the private sector in Turkey
* For senior students studying in the physiotherapy and rehabilitation department
* Volunteer to participate in the study

Exclusion Criteria:

* Not to be a physiotherapist
* Those who study in the physiotherapy and rehabilitation department but are not final year students
* Not volunteering to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapists working in various institutions and the private sector in Turkey and senior students studying in the physiotherapy and rehabilitation department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level of Cardiopulmonary Resuscitation | 5 months
  Cardiopulmonary resuscitation knowledge level survey result

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Tugba Kilic, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Result] Travers AH, Rea TD, Bobrow BJ, Edelson DP, Berg RA, Sayre MR, Berg MD, Chameides L, O'Connor RE, Swor RA. Part 4: CPR overview: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S676-84. doi: 10.1161/CIRCULATIONAHA.110.970913. No abstract available. PMID 20956220
- [Result] Sandroni C, Nolan J; European Resuscitation Council. ERC 2010 guidelines for adult and pediatric resuscitation: summary of major changes. Minerva Anestesiol. 2011 Feb;77(2):220-6. PMID 21368728
- [Result] Schneider AP 2nd, Nelson DJ, Brown DD. In-hospital cardiopulmonary resuscitation: a 30-year review. J Am Board Fam Pract. 1993 Mar-Apr;6(2):91-101. PMID 8452077
- [Result] Kiyan S, Yanturali S, Musal B, Gursel Y, Aksay E, Turkcuer I. Determination of advanced life support knowledge level of residents in a Turkish university hospital. J Emerg Med. 2008 Aug;35(2):213-22. doi: 10.1016/j.jemermed.2007.02.049. Epub 2007 Jul 20. PMID 17976765
- [Result] Jonathon Webber R. Knowledge and perceptions of cardiopulmonary resuscitation amongst New Zealand physiotherapists. New Zealand Journal of Physiotherapy. 2019;47(2):94-104.
- [Result] Mbada CE, Hakeem BO, Adedoyin RA, Awotidebe TO, Okonji AM. Knowledge, attitude and practive of cardiopulmonary resuscitation among Nigerian physiotherapists. Journal of Respiratory and Cardiovascular Physical Therapy. 2013;2(2):52-62.